CLINICAL TRIAL: NCT07183865
Title: Hypofractionated Radiotherapy Combined With Irinotecan Hydrochloride Liposome, 5-FU, Leucovorin, PD-1 Antibody and Target Therapy in Locally Recurrent Rectal Cancer(NOVELTY-R)
Brief Title: Hypofractionated Radiotherapy Combined With NALIRIF, PD-1 Antibody in Locally Recurrent Rectal Cancer(NOVELTY-R)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Department of Radiation Oncology, Fudan University Shanghai Cancer Center, Shanghai, China, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-383-3937
Record Dates: First submitted 2025-04-08; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Locally Recurrent Rectal Cancer
MeSH Terms: interventions — Radiotherapy; Fluorouracil; Leucovorin; Cetuximab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Radiotherapy:
  The enrolled patients will receive 25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation (pelvic radiation history) for pelvic recurrence.All metastasis sites will receive 25-50Gy/5Fx irradiation before or between system therapy cycles. Dose Constraints are based on SABR-COMET 10 trial.
  System therapy:
  Patients will receive Irinotecan Hydrochloride Liposome plus 5-FU and leucovorin (NALIRIF), PD-1 antibody, target therapy based on the KRAS/NRAS/BRAF mutation station.
  Interventions: Radiation: radiotherapy; Drug: Irinotecan Hydrochloride Liposome; Drug: 5-FU; Drug: Leucovorin; Drug: SG001; Drug: C225; Drug: Bevacizumab

INTERVENTIONS:
Radiation: radiotherapy — 25-40Gy/5Fx or 15-30Gy/5Fx (previous pelvic radiation) for pelvic recurrence. 25-50GY/5Fx for all metastasis tumors. Dose Constraints are based on SABR-COMET 10 trial.
Drug: Irinotecan Hydrochloride Liposome — 70mg/m2 (UGT1A1*28 6/6) or 55mg/m2 (UGT1A1*28 6/7), IV, q2w
Drug: 5-FU — 400 mg/m^2 bolus over 2 hours followed by 2400 mg/m^2 continuous infusion over 48 hours d1, q2w
Drug: Leucovorin — 400mg/m2, IV, q2w
Drug: SG001 — 240mg, IV, q2w
Drug: C225 — 500 mg/m2, IV, q2w
Drug: Bevacizumab — 5mg/kg, IV, q2w

SUMMARY:
This is an open-label, single arm, phase 2 study. The study is to evaluate the activity of combination therapy of hypofractionated radiotherapy, Irinotecan Hydrochloride Liposome plus 5-FU and leucovorin (NALIRIF), Anti-PD1 and target therapy in patients with locally recurrent rectal cancer (LRRC). The inclusion LRRC patients were failed to oxaliplatin treatment in prior chemotherapy or chemoradiotherapy due to toxicity or progression. Patients will receive 25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation for pelvic recurrence, 25-50Gy/5Fx irradiation for all metastasis sites, and 8 cycles of NALIRIF + anti-PD1 + target therapy, followed by multidisciplinary team (MDT) for decision: radical surgery, sustained system +/- local treatment of non resection.

The primary endpoint was local objective response rate. Secondary endpoints were extrapelvic objective response rate, complete response rate, R0 resection rate, duration of response, progression-free survival, overall survival, and safety and tolerability of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Patient is 18-75 years old at the time of signing the informed consent form. ECOG performance status 0-1. MRI/enhanced CT confirmed pelvic recurrence. According to RECIST 1.1, there is at least one measurable pelvic lesion.

Distant metastasis lesions are no more than 5 and metastatic organ are no more than 3.

No prior radiotherapy within 6 month. Failed to oxaliplatin treatment in prior chemotherapy or chemoradiotherapy due to toxicity or progression.

Has an investigator determined life expectancy of at least 24 weeks. Demonstrate adequate organ function (bone marrow, liver, kidney and clotting function) within 7 days before the first administration without using blood products or hematopoietic stimulating factors.

Non pregnant or lactating patients. Effective contraceptive methods should be used during the study and within 6 months of the last administration.

Fully informed and willing to provide written informed consent for the trial.

Exclusion Criteria:

Previous immunotherapy or Irinotecan Hydrochloride Liposome treatment. Neutrophil < 1.5×10^9/L, PLT < 100×10^9/L (PLT < 80×10^9/L in patients with liver metastasis), or Hb < 90g/L; blood transfusion within 2 weeks before enrollment is not allowed to meet the enrollment criteria.

TBIL > 1.5 ULN, or TBIL > 2.5 ULN in patients with liver metastasis. AST or ALT > 2.5 ULN, or ALT and / or AST > 5 ULN in patients with liver metastasis.

Cr > 1.5 ULN, or creatinine clearance < 50ml / min (calculated according to Cockcroft Gault formula).

APTT > 1.5 ULN, PT > 1.5 ULN (subject to the normal value of the clinical trial research center).

Serious electrolyte abnormalities. Urinary protein ≥ 2+, or 24-hour urine protein ≥1.0g/24h. Uncontrolled hypertension: SBP >140mmHg or DBP > 90mmHg. The presence of gastrointestinal diseases such as gastric or duodenal active ulcers, ulcerative colitis or unresected tumours with active bleeding; or other conditions likely to cause gastrointestinal bleeding or perforation; or unhealed gastrointestinal perforation or gastrointestinal fistula after surgical treatment.

A history of arterial thrombosis or deep vein thrombosis within 6 months; a history of bleeding or evidence of bleeding tendency within 2 months.

A history of heart disease within 6 months (including congestive heart failure, acute myocardial infarction, severe/unstable angina, coronary artery bypass grafting, cardiac insufficiency ≥ NYHA grade 2 and LVEF<50%).

Uncontrolled malignant pleural effusion, ascites, or pericardial effusion. The presence of a clinically detectable second primary malignancy, or history of other malignancies within 5 years excluding adequately treated non-melanoma skin cancer, carcinoma in situ of cervix and superficial bladder tumour (non-invasive tumour, or carcinoma in situ, or T1).

A history of liver disease including, but not limited to HBV infection or HBV DNA positive(≥1×10^4/ml), HCV infection or HCV DNA positive(≥1×10^3/ml) and liver cirrhosis.

Pregnant or lactating women or women who may be pregnant have a positive pregnancy test before the first medication; Or the female participants themselves and their partners who were unwilling to implement strict contraception during the study period.

The investigator considers that the subject is not suitable to participate in this clinical study due to any clinical or laboratory abnormalities or compliance problems.

Serious mental abnormalities. The diameter of brain metastasis is greater than 3cm or the total volume is greater than 30cc.

Clinical or radiological evidence of spinal cord compression, or tumours within 3 mm of the spinal cord on MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2030-03-09 (Estimated); Study Completion 2030-03-09 (Estimated)

PRIMARY OUTCOMES:
Local objective response rate | up to 1 year
  the proportion of patients with the best pelvic response of confirmed complete or partial response according to RECIST 1.1, as assessed by the investigator.

SECONDARY OUTCOMES:
Extrapelvic objective response rate | up to 1 year
  proportion of patients with confirmed extrapelvic complete or partial response per RECIST 1.1.
Complete response rate | up to 1 year
  proportion of patients with confirmed complete response per RECIST 1.1.
R0 resection rate | up to 1 year
  the proportion of patients who achieve R0 resection of pelvic recurrent tumour after therapy.
Duration of response (DOR) | up to 3 year
  time from the first documented pelvic objective response to pelvic or extrapelvic disease progression in patients with confirmed response.
Progression-Free Survival(PFS) | up to 3 year
  time from the date of start treatment until disease progression or censored at last follow-up or death.
Overall Survival | up to 3 year
  from the date of start treatment until the date of death from any cause or censored at last follow-up.
Safety and tolerability of the treatment | up to 1 year
  proportion of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China